CLINICAL TRIAL: NCT01942109
Title: The Impact of TORasemide oN hemodynAmic and Neurohormonal Stress, and carDiac remOdeling in Heart Failure - Prospective, Randomized, Open, Blinded Endpoint Trial
Brief Title: The Impact of TORasemide oN hemodynAmic and Neurohormonal Stress, and carDiac remOdeling in Heart Failure
Acronym: TORNADO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TORNADO KB/202/2013
Record Dates: First submitted 2013-08-24; First posted 2013-09-13 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
Keywords: heart failure; diuretics; furosemide; torasemide
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Torsemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide (Active Comparator): This group will receive furosemide as a diuretic treatment
  Interventions: Drug: Furosemide
- Torasemide (Experimental): This group will receive torasemide as a diuretic treatment
  Interventions: Drug: Torasemide

INTERVENTIONS:
Drug: Furosemide — Drug will be administered per os. Dose of the agent will be adapted to clinical status of the patient. Equipotential dose for furosemide is torasemide in dose 1:4 of furosemide
  Arms: Furosemide
Drug: Torasemide — Drug will be administered per os. Dose of the agent will be adapted to clinical status of the patient. Equipotential dose for furosemide is torasemide in dose 1:4 of furosemide
  Arms: Torasemide

SUMMARY:
The aim of the study is to compare the effects of torasemide and furosemide on clinical and biochemical parameters of hemodynamic and neurohormonal compensation and myocardial remodeling in patients with chronic heart failure with indications for use of loop diuretics.

The study protocol 100 patients with heart failure NYHA (New York Heart Association) II-IV (stable or exacerbation aligned cardiopulmonary at the time of enrollment, with a fixed-dose loop diuretics]) treated with optimal medical therapy as clinically indicated for use loop diuretics. Patients will be randomized to treatment with furosemide and torasemide (randomization 1 : 1). After randomization, furosemide will continue in its current fixed-dose or will be replaced by equipotential dose of torasemide (4:1). The minimal follow-up of patients in the study will be at least six months.

DETAILED DESCRIPTION:
According to current guidelines, angiotensin converting enzyme inhibitors and beta-adrenolytics are the first-line treatment agents in patients with heart failure. In case of fluid retention, diuretics, as a part of symptomatic treatment, should be administered. In practice, the most common diuretic used in patients with heart failure is loop diuretic - furosemide. What is important, furosemide has no effect on patients' outcomes. Some studies showed unfavourable influence of this drug on rennin-angiotensin-aldosterone system.

Alternative loop diuretic, which may be administered in patients with heart failure is torasemide. Its longer elimination half-life time, similar diuretic effects, lower influence on electrolyte disorders and additional pleiotropic effects could make torasemide more beneficial than furosemide.

Accordingly, only direct comparison of furosemide and torasemide could present similarities and differences of these two agents.

The hypothesis of this study is that torasemide may present more favourable effects on some clinical parameters in patients with heart failure, than furosemide (e.g. clinical symptoms, biochemical parameters, activity of rennin-angiotensin-aldosterone system, side effects).

ELIGIBILITY:
Inclusion Criteria:

* heart failure NYHA II-IV
* previous treatment with diuretics
* age>18 years

Exclusion Criteria:

* uncontrolled hypertension
* uncontrolled diabetes
* creatinine > 2,5 mg/dl
* potassium > 6 mg/dl
* acute coronary syndrome
* hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The influence of therapy on cardiovascular events associated with heart failure (deaths, hospitalisations) | up to 12 months

SECONDARY OUTCOMES:
The change of dosing of diuretic due to worsening of condition of patient. | up to 12 months
The change of NYHA (New York Heart Association) class - worsening or improvement | up to 12 months

OTHER OUTCOMES:
The measurement of fluid retention with ZOE Fluid Status Monitor | up to 12 months
≥30% or ≥200 pg/ml increase of NTproBNP (N-terminal pro B type natriuretic peptide) level compared with baseline value | up to 12 months
The change between baseline and final levels of serum biomarkers | up to 12 months
The assessment of quality of life | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Grabowski, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw
Locations (2):
- Poland (2):
  - 3rd Clinic of Internal Medicine and Cardiology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship
  - 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship

REFERENCES:
- [Derived] Balsam P, Ozieranski K, Tyminska A, Glowczynska R, Peller M, Fojt A, Cacko A, Sieradzki B, Bakula E, Markulis M, Kowalik R, Huczek Z, Filipiak KJ, Opolski G, Grabowski M. The impact of torasemide on haemodynamic and neurohormonal stress, and cardiac remodelling in heart failure - TORNADO: a study protocol for a randomized controlled trial. Trials. 2017 Jan 23;18(1):36. doi: 10.1186/s13063-016-1760-z. PMID 28114980